CLINICAL TRIAL: NCT02436421
Title: Impact of Best Practice Alerts in Cardiology Outpatient Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00045379
Record Dates: First submitted 2015-05-04; First posted 2015-05-06 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension; Atrial Fibrillation
MeSH Terms: conditions — Hypertension; Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atrial Fibrillation BPA (Other): The alert will notify providers when patients with atrial fibrillation are not on anticoagulation
  Interventions: Other: Best Practice Alert based in the Electronic Medical Record
- Hypertension BPA (Other): The alert will notify providers when patients have elevated blood pressure
  Interventions: Other: Best Practice Alert based in the Electronic Medical Record
- Atrial Fibrillation and Hypertension BPA (Other): Providers in this arm will receive both alerts
  Interventions: Other: Best Practice Alert based in the Electronic Medical Record

INTERVENTIONS:
Other: Best Practice Alert based in the Electronic Medical Record

SUMMARY:
This quality improvement intervention seeks to implement two Best Practice Alerts (BPAs) for use in cardiology clinics while simultaneously evaluating the impact of each BPA- one for patients with uncontrolled blood pressure and one for patients with atrial fibrillation not on anticoagulation.

DETAILED DESCRIPTION:
Best Practice Alerts based will be created for hypertension and atrial fibrillation. Outpatient cardiology providers will be randomly allocated into one of three groups. The first group will receive the BPA for hypertension alone. The second group will receive the BPA for atrial fibrillation alone. The final group will receive both BPAs. The rate of blood pressure control for all patients and anticoagulation in patients with atrial fibrillation in each group will be evaluated prior to and after the implementation of the BPAs to determine the effect of the BPA.

ELIGIBILITY:
Inclusion Criteria:

* all patients seen routinely by cardiologists at Duke

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Rates of anticoagulation among patients with atrial fibrillation | 1 year
Rates of hypertension control among patients seen by cardiology | 1 year